CLINICAL TRIAL: NCT07170033
Title: A New Approach to Nutritional Therapy in Rheumatoid Arthritis: Evaluation of the Effect of the DASH Diet Through a Randomized Controlled Clinical Trial
Brief Title: The Effect of the DASH Diet on Treatment Outcomes in Adults Diagnosed With Rheumatoid Arthritis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Health and Technology University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Gokcen Ozupek, PhD Candidate, Istanbul Health and Technology University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ISTUN-GO-01
Record Dates: First submitted 2025-09-07; First posted 2025-09-12 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Rheumatoid Arthritis
Keywords: Diet Therapy; Inflammation; Dietary Approaches To Stop Hypertension; Randomized Controlled Trial
MeSH Terms: conditions — Arthritis, Rheumatoid; Inflammation | interventions — Diet

STUDY DESIGN:
Intervention Model Description: This is a randomized, controlled, parallel-group trial in which participants diagnosed with seropositive rheumatoid arthritis will be assigned to either a DASH diet intervention group or a control group maintaining their habitual dietary intake. The study duration is 12 weeks.
Masking Description: This is an open-label study. No masking was applied, as both participants and investigators were aware of the group assignments due to the nature of the dietary intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DASH Diet Group (Experimental): Participants in this group will follow the DASH diet for 12 weeks. The diet will be tailored according to individual physical activity levels and basal metabolic rate. Dietary adherence will be monitored through dietary intake records and DASH diet scores calculated using the Nutrition Information System (BeBiS).
  Interventions: Other: Dietary Approach to Stop Hypertension (DASH) Diet
- Control Group (No Intervention): Participants in this group will continue their usual diet without any dietary intervention. They will be monitored for the same outcomes as the intervention group during the 12-week study period.

INTERVENTIONS:
Other: Dietary Approach to Stop Hypertension (DASH) Diet — "Dietary intervention: DASH diet" Participants in the intervention group will follow the Dietary Approaches to Stop Hypertension (DASH) diet for 12 weeks. The diet plan will be personalized based on each participant's 24-hour physical activity level and basal metabolic rate. Dietary adherence will be monitored through 3-day dietary intake records and DASH diet scores calculated using the Nutrition Information System (BeBiS). The intervention aims to assess the effect of the DASH diet on inflammatory markers, disease activity scores, functional status, and quality of life in adults diagnosed with seropositive rheumatoid arthritis.
  Arms: DASH Diet Group

SUMMARY:
In this study, it is aimed to determine the effect of the DASH diet model on the treatment of patients with seropositive rheumatoid arthritis, by evaluating its potential impact on inflammatory markers, disease activity scores, patients' functional status in daily life, and quality of life.

"This study is being conducted as part of a doctoral dissertation, and due to insufficient initial awareness regarding the requirement for prior registration, the registration process was completed after data collection had already begun. However, data collection is still ongoing, and the study has not yet been completed. We remain committed to full compliance with clinical trial reporting standards and transparency."

DETAILED DESCRIPTION:
Prior to the commencement of the study, participants will be informed about the research, and those who voluntarily agree to participate will be asked to sign an informed consent form. This study, designed to determine the effect of the DASH diet on treatment outcomes in patients diagnosed with seropositive rheumatoid arthritis (RA), will collect data through a questionnaire including participants' demographic characteristics (gender, age, marital status, education level, occupation, income status), health status (duration of treatment, RA symptoms, presence of RA in relatives, use of medications and nutritional supplements, history of any RA-specific nutritional or diet therapy, presence of any chronic diseases other than RA, pregnancy/lactation status in RA patients), dietary habits (number of main and snack meals, reasons for meal skipping, foods consumed during snacks, average daily water intake, smoking and alcohol consumption), functional status in daily life, quality of life, food consumption frequency, and a 3-day dietary record. Additionally, numerical data including patients' 24-hour physical activity level, DAS-28 disease activity score, VAS general health assessment, VAS pain score, anthropometric measurements (body weight, height, and BMI), and basal metabolic rate (BMR) will be obtained.The DASH diet prescribed to patients in the intervention group will be planned according to their 24-hour physical activity level and BMR. The DASH diet adherence score will be calculated using the "Nutrition Information System (BeBiS)" program, based on the patients' dietary intake records including average daily intake of total fat, saturated fat, protein, cholesterol, fiber, magnesium, calcium, sodium, and potassium. Biochemical findings of the patients will be obtained from the patient information system with physician approval.This randomized controlled trial is planned to implement the DASH diet intervention for 3 months (12 weeks), considering similar studies in the literature, to observe the expected differences in patients with seropositive rheumatoid arthritis in the intervention group. Patients in the control group will continue their usual diet without any specific dietary intervention. Relevant data from individuals in both the intervention and control groups will be collected again at the end of weeks 4, 8, and 12 following the dietary intervention.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary acceptance to participate in the study, Being within the age range of 18-64 years, Having a diagnosis of rheumatoid arthritis according to the 2010 American College of Rheumatology (ACR)/European League Against Rheumatism (EULAR) classification criteria and belonging to the seropositive rheumatoid arthritis subgroup, Being in the active phase of rheumatoid arthritis according to the DAS-28 CRP or DAS-28 ESR disease activity score, Having a disease duration of at least 1 year, Not having previously undergone any dietary treatment specific to rheumatoid arthritis, Not using any dietary supplements other than calcium and vitamin D3 supplementation (e.g., 1000 mg calcium, 880 IU vitamin D3) recommended by the physician for patients using glucocorticoids and folic acid supplementation (10 mg weekly) recommended for patients using methotrexate, Having stable use of disease-modifying anti-rheumatic drugs (≥3 months), corticosteroids (≥4 weeks), and nonsteroidal anti-inflammatory drugs (≥10 days) before starting the DASH diet treatment, with a daily oral corticosteroid dose not exceeding 12.5 mg of prednisolone, Not having a diagnosis of eating disorders, Not being pregnant or breastfeeding, Not using banned substances, Having no intellectual disability, Having no allergy and/or intolerance to the foods included in the DASH diet

Exclusion Criteria:

* Not voluntarily agreeing to participate in the study, Not being within the age range of 18-64 years, Not having a diagnosis of rheumatoid arthritis according to the 2010 American College of Rheumatology (ACR)/European League Against Rheumatism (EULAR) classification criteria, and not belonging to the seropositive rheumatoid arthritis subgroup, Being in remission according to the DAS-28 CRP and DAS-28 ESR disease activity scores, Having a disease duration of less than 1 year, Having previously undergone any dietary treatment specific to rheumatoid arthritis, Using any dietary supplements other than calcium and vitamin D3 supplementation (e.g., 1000 mg calcium, 880 IU vitamin D3) recommended by the physician for patients receiving glucocorticoid therapy and folic acid supplementation (10 mg weekly) recommended for patients using methotrexate, Having changes in disease-modifying anti-rheumatic drugs usage within less than 3 months, corticosteroids within less than 4 weeks, and nonsteroidal anti-inflammatory drugs within less than 10 days before starting the DASH diet treatment, having a daily oral corticosteroid dose exceeding 12.5 mg of prednisolone, Having a diagnosis of eating disorders, Being pregnant or breastfeeding, Using banned substances, Having intellectual disability, Having any allergy and/or intolerance to the foods included in the DASH diet.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2024-05-06 (Actual); Primary Completion 2025-10-06 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in Disease Activity Score-28 (DAS-28) | Baseline, Week 4, Week 8, and Week 12
  Disease activity will be assessed using the Disease Activity Score-28 (DAS-28), calculated with both C-reactive protein (CRP) and erythrocyte sedimentation rate (ESR). DAS-28 scores will be recorded at baseline, and at Weeks 4, 8, and 12. The change over time will be used to evaluate the effectiveness of the DASH diet intervention in patients with rheumatoid arthritis. According to the calculated DAS-28 score, a value of ≤3.2 indicates low disease activity; a score between >3.2 and ≤5.1 indicates moderate disease activity; and a score >5.1 indicates high disease activity. A DAS-28 score of <2.6 is defined as remission.

SECONDARY OUTCOMES:
Change in Pain Score Measured by Visual Analog Scale (VAS) | Baseline, Week 4, Week 8, and Week 12
  Pain intensity will be assessed using the Visual Analog Scale (VAS), which ranges from 0 (no pain) to 10 (worst possible pain). The change in VAS pain scores will be recorded at baseline, Week 4, Week 8, and Week 12 to evaluate the effect of the DASH diet intervention on pain levels in patients with rheumatoid arthritis. Pain intensity is classified as mild for scores <3; moderate for scores between 3 and 6; and severe for scores >6.
Change in Biochemical Parameters | Baseline, Week 4, Week 8, and Week 12
  Changes in biochemical parameters (such as inflammatory markers including CRP and ESR) will be monitored at baseline, Week 4, Week 8, and Week 12 to evaluate the biochemical response to the DASH diet intervention in patients with rheumatoid arthritis.
Change in Scores from Health Assessment Questionnaire | Baseline, Week 4, Week 8, and Week 12
  Scores obtained from the Health Assessment Questionnaire (HAQ) will be recorded at baseline, Week 4, Week 8, and Week 12 to assess changes in patients' functional status and overall health following the DASH diet intervention. The scale score ranges from 0 to 3, with higher scores indicating poorer health status.
Change in Scores from the Short Form-36 (SF-36) Health Survey | Baseline, Week 4, Week 8, and Week 12
  Scores obtained from the Short Form-36 (SF-36) Health Survey will be recorded at baseline, Week 4, Week 8, and Week 12 in patients with rheumatoid arthritis to evaluate changes in quality of life. An increase in the scores on the scale indicates an improvement in health-related quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Gökçen ÖZÜPEK, Principal Investigator — Istanbul Health and Technology University; İkbal S ALTAY, AsstProf, Study Chair — Istanbul Health and Technology University; Zeynep B KALYONCU ATASOY, AsstProf, Study Director — Saglik Bilimleri Universitesi
Locations (2):
- Turkey (Türkiye) (2):
  - Başakşehir Çam and Sakura City Hospital, Istanbul
  - Istanbul Prof. Dr. Cemil Taşcıoğlu City Hospital, Istanbul

IPD SHARING:
Plan to Share IPD: No